CLINICAL TRIAL: NCT03631420
Title: The Safety and Feasibility of UMC119-01 Cell Therapy in Infants at High Risk for Bronchopulmonary Dysplasia
Brief Title: Mesenchymal Stem Cells for Prevention of Bronchopulmonary Dysplasia in Infants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Meridigen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMC119-01-001
Record Dates: First submitted 2018-04-09; First posted 2018-08-15 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-12

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UMC119-01 (Experimental): UMC119-01 is ex vivo cultured human umbilical cord tissue-derived mensenchymal stem cells product
  Interventions: Biological: Human Umbilical Cord Derived-Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Human Umbilical Cord Derived-Mesenchymal Stem Cells — Cohort 1 : 3 million cells/kg ; Cohort 2 : 10 million cells/kg ; Cohort 3 : 30 million cells/kg

SUMMARY:
The clinical study with UMC119-01 is designed to investigate the safety in patients with bronchopulmonary dysplasia ("BPD"). This will be a dose escalation, open-label, single-center study in infants at high risk for BPD.

DETAILED DESCRIPTION:
UMC119-01 is ex vivo cultured human umbilical cord tissue-derived mensenchymal stem cells product which is intended for prevention of Bronchopulmonary dysplasia.

ELIGIBILITY:
Inclusion Criteria:

Neonatal infants who fulfil all of the following criteria will be enrolled:

1. Subjects of postnatal age between 3 to 30 days.
2. Are male and female infants born at GA between 23 weeks to 29 weeks. The postmenstrual age of subject received UMC119-01 should be no more than PMA36 weeks.
3. Subjects with birth weight between 501g to 1249 g.
4. Have endotracheal tube in place as part of SoC for preterm infants with BPD at screening and on treatment visit (Day 0), and that they will have not been intubated for the purposes of this study.
5. A subject who is intubated and receiving mechanical ventilation with a fraction of inspired oxygen (FiO2) of 0.25 or greater at Screening.
6. A subject who has had either a deterioration or no change in the setting of mechanical ventilation within the 24 hours before trial enrollment.
7. Written informed consent has been provided by the subject's parents, legal guardians, or a legal representative, who agree to comply with all of the study procedures, including those in the long-term safety surveillance period.

Exclusion Criteria:

Neonatal infants who meet any of the following criteria will be excluded:

1. Have a major congenital abnormality, including neurological (including anencephaly and similar malformations), hepatic, renal, cardiovascular abnormality (except for patent ductus arteriosus, PDA).
2. Have a known genetic syndrome.
3. Have a condition that makes them ineligible for participation in this study, as determined by the investigator.
4. Have C-reactive protein (CRP) >30 mg/L; or any infections including pneumonia, sepsis, or shock.
5. Have pre-existing severe intraventricular hemorrhage (IVH) (grade ≥3).
6. Have active pulmonary hemorrhage or air leak syndrome.
7. Have abnormal hepatic (AST, ALT >150 U/L or direct bilirubin >2 mg/dL or total bilirubin >15 mg/dL) or renal function (serum creatinine >1 mg/dL or oliguria).
8. Are known to be infected with HIV or CMV.
9. Are expected to have surgery within 24 hours prior to and/or after UMC119 01 instillation.
10. Are expected to receive any other intratracheal treatments, including surfactant within 72 hours prior to and/or after UMC119 01 instillation.
11. Are currently participating in any other interventional clinical trial.

Ages: 3 Days to 51 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of adverse events related to administration of UMC119-01. | 3 months from the day of administration
  • The incidence and frequency of adverse events (AEs) and serious adverse events (SAEs), including their relationship to the administration of UMC119 01.

SECONDARY OUTCOMES:
The percentage of subjects who died from any cause during the study. | 3 months from the day of administration
  The percentage of subjects who died from any cause during the study.
Changes of the oxygen saturation. | 3 months from the day of administration
  Changes from baseline of the oxygen saturation.
Changes of chest x-ray findings in participants before and after administration. | 3 months from the day of administration
  Changes from baseline to 3 months of chest x-ray findings in participants before and after administration.
Changes of inflammatory markers (pg/ml) before and after administration. | 3 days and 7 days after administration
  Changes from baseline of inflammatory markers (pg/ml) .
Comparison of the incidence and severity of preterm children's complications in participants before and after administration. | 3 months from the day of administration
  Comparison of the incidence and severity of preterm children's complications in participants before and after administration.
The number of days of intubation, or where ventilator or oxygen therapy. | 3 months from the day of administration
  The number of days of intubation, or where ventilator or oxygen therapy.
Incidence of moderate/severe BPD or death at 36 weeks postmenstrual age (PMA). | 36 weeks postmenstrual age (PMA)
  Incidence of moderate/severe BPD or death at 36 weeks postmenstrual age (PMA).

CONTACTS AND LOCATIONS:
Locations (1):
- National Chen-Kung University Hospital, Tainan, Taiwan